CLINICAL TRIAL: NCT00102427
Title: Improving Quality of Primary Care for Anxiety Disorders
Brief Title: Improving Quality of Primary Care for Patients With Anxiety and/or Panic Disorders
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH059395 (NIH); R01MH059395 (NIH)
Record Dates: First submitted 2005-01-29; First posted 2005-01-31 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Panic Disorder; Anxiety Disorder
Keywords: Anxiety; Panic; Generalized Anxiety Disorder
MeSH Terms: conditions — Panic Disorder; Anxiety Disorders; Generalized Anxiety Disorder

INTERVENTIONS:
Behavioral: Telephone-based collaborative care management

SUMMARY:
The purpose of this study is to determine if primary care patients with panic and/or generalized anxiety disorder can benefit from a telephone-based collaborative care intervention.

DETAILED DESCRIPTION:
Panic and generalized anxiety disorders are serious conditions that often are inadequately recognized and treated, responsible for significant morbidity, and associated with excessive health services' utilization. More effective treatment interventions that involve both primary care physicians (PCPs) and patients are necessary to manage these conditions.

Patients presenting for primary care services will be screened for panic and generalized anxiety disorders using the Primary Care Evaluation of Mental Disorder (PRIME-MD); patients and their PCPs will be informed of patients' diagnosis. Participants will then be randomly assigned to receive either a telephone-based collaborative care intervention or their PCPs' usual care.

The telephone care intervention will involve a protocol that is based on the American Psychiatric Association's and other published guidelines for treating panic disorder (PD) and generalized anxiety disorder (GAD). The care manager will assess each patient's treatment preferences for either anxiolytic pharmacotherapy, a self-management workbook, referral to a community mental health specialist, or some combination of these. The care manager will conduct periodic telephone follow-up interviews with intervention participants to inquire about anxiety symptoms, treatment adherence, review lesson plans, and any side effects they have experienced, as applicable. The care manager maintains correspondence with the PCPs of the telephone intervention participants via an electronic medical record system to rapidly relay information regarding patients' treatment and obtain the PCPs approval for initiating or adjusting pharmacotherapy according to the patient's response to treatment and protocol.

A blinded research assistant who is unaware of participants' randomization group will conduct telephone interviews with all participants to assess the effectiveness of the intervention relative to the usual care control condition. These interviews will be conducted at baseline and at 2-, 4-, 8-, and 12-months follow-up. Measures assessed include anxiety symptoms, functional status, health services utilization, and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Panic disorder or generalized anxiety disorder
* A Structured Interview Guide to the Hamilton Rating Scale for Anxiety (SIGH-A) score of at least 14 for participants with generalized anxiety disorder OR Panic Disorder Severity Scale (PDSS) score of at least 7 for participants with panic disorder
* Primary care physician has agreed to participate in the study
* Speaks English and able to participate in phone assessments and information/self-management program
* Gives consent to allow research staff to notify the participant's primary care physician of diagnosis

Exclusion Criteria:

* Thoughts of suicide
* Current psychotic disorder
* Current bipolar disorder
* Alcohol or other substance disorder within the past 2 months prior to study entry
* Organic anxiety syndromes, including those due to medical illness or drugs
* Unstable medical conditions
* Plans to leave current physician during the year after study start
* Life expectancy less than 1 year
* Previously enrolled in a similar panic or generalized anxiety disorder study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2000-07; Study Completion 2003-05

PRIMARY OUTCOMES:
Anxiety symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Bruce L. Rollman, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Rollman BL, Herbeck Belnap B, Reynolds CF, Schulberg HC, Shear MK. A contemporary protocol to assist primary care physicians in the treatment of panic and generalized anxiety disorders. Gen Hosp Psychiatry. 2003 Mar-Apr;25(2):74-82. doi: 10.1016/s0163-8343(03)00004-5. PMID 12676419
- [Result] Rollman BL, Belnap BH, Mazumdar S, Houck PR, Zhu F, Gardner W, Reynolds CF 3rd, Schulberg HC, Shear MK. A randomized trial to improve the quality of treatment for panic and generalized anxiety disorders in primary care. Arch Gen Psychiatry. 2005 Dec;62(12):1332-41. doi: 10.1001/archpsyc.62.12.1332. PMID 16330721
- [Derived] Rollman BL, Fischer GS, Zhu F, Belnap BH. Comparison of electronic physician prompts versus waitroom case-finding on clinical trial enrollment. J Gen Intern Med. 2008 Apr;23(4):447-50. doi: 10.1007/s11606-007-0449-0. PMID 18373143